CLINICAL TRIAL: NCT04372719
Title: An Open-Label, Ascending Dose Study to Determine the Safety and Attack Rate of a Wild Type, Seasonal H3N2 Influenza Challenge Agent in Healthy Volunteers
Brief Title: A Study to Determine the Safety and Attack Rate of the Seasonal Flu in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHAMP-H3N2
Record Dates: First submitted 2020-04-22; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H3N2 10EXP5 TCID50/mL (Experimental): A/Belgium/4217/2015 (H3N2) (SGS Code: SGS 421-7), Wild-type, influenza A (H3N2) human challenge strain
  Interventions: Drug: H3N2

INTERVENTIONS:
Drug: H3N2

SUMMARY:
This is a non-controlled, open-label, single-centre, dose-escalation study to determine the safety, infectivity and immunology of the potential novel influenza virus H3N2 challenge strain. The term 'challenge agent' used in this protocol refers to the Influenza virus H3N2 A/Belgium/4217/2015. The study utilises an adaptive study design and consists of 2 parts.

DETAILED DESCRIPTION:
In Part 1, the primary objective is to determine the viral challenge strain dose that has an acceptable safety profile and an observed attack rate of >60% (i.e., at least 8 out of 12 subjects should be infected). After Part 1, a formal interim analysis will be performed to select the viral challenge strain dose for Part 2 by evaluating the primary objective of Part 1. In case no viral challenge strain dose can be selected, the study will not proceed to Part 2.

In Part 2, the primary objective is to determine the infectivity rate in healthy volunteers of the selected viral challenge strain dose for use in subsequent human challenge intervention studies.

All subjects will be screened prior to viral inoculation to assess their suitability to enter the study. Eligible subjects will be admitted to the clinical centre for a single intranasal inoculation with influenza A (H3N2). In this study, up to 64 healthy subjects will receive the investigational challenge agent: 36 subjects in Part 1 and 18 or 28 subjects in Part 2.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, between 18 and 55 years old (extremes included) at screening.
2. In good physical and mental health as determined on the basis of medical history and general physical examination performed at screening.
3. Absent or low levels of detectable pre-existing antibodies to influenza virus subtypes, including as a minimum the challenge strain, as determined by a MNT titre of ≤ 20 at screening.
4. Negative urine test for selected drugs of abuse at screening and upon check-in at the clinical site.
5. Negative alcohol breath test
6. Female subjects should fulfil one of the following criteria:

   1. At least 1 year post-menopausal (amenorrhea >12 months and/or follicle-stimulating hormone (FSH) > 30 mIU/mL) prior to screening;
   2. Surgically sterile (bilateral oophorectomy, hysterectomy, or tubal ligation);
   3. Will use contraceptives as outlined in inclusion criterion 8 from screening to discharge.
7. Female subjects of childbearing potential and male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control from screening to discharge.

Exclusion criteria:

1. Subjects who have received any vaccination within the last 3 months prior to screening or influenza vaccine within the last 12 months prior to screening or who anticipate receiving this during the study.
2. Subjects with a diagnosis of influenza or influenza-like illness confirmed by a physician within the last 6 months prior to screening.
3. Subjects with a positive result for adventitious agent screening (qualitative PCR testing) for any respiratory virus or bacteria on Day -2.
4. Haematology and chemistry parameters, pulse rate and/or blood pressure, and ECG outside the reference range for the population studied and considered as clinical significant by the Investigator.
5. Has an acute or chronic medical condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
safety profile | through study completion, an average of 3 months
  Number of subjects with SAEs considered by the Investigator to be related to the challenge agent, moderate or severe lower respiratory symptoms as indicated on the symptom score card, or confirmed cytokine-related AEs.
Efficacy: Infectivity | through study completion, an average of 3 months
  Attack rate defined as number of inoculated subjects with any of the following:
  * Fever
  * At least one other (i.e., not fever) influenza symptom At least 2 consecutive swabs positive for H3N2
Efficacy: observed attack rate | through study completion, an average of 3 months
  Observed attack rate expressed in percentage

SECONDARY OUTCOMES:
Safety: Incidence of Related virus-emergent adverse events | through study completion, an average of 1 year
  Safety: Incidence of Related virus-emergent adverse events

IPD SHARING:
Plan to Share IPD: No